CLINICAL TRIAL: NCT02594800
Title: The Impact of Intensive Rosuvastatin Therapy on Cerebral Hemodynamics in Patients With Atherosclerotic Intracranial Arterial Stenosis Evaluated by Computed Tomography Perfusion (CTP)
Brief Title: Intensive Rosuvastatin Therapy on Cerebral Hemodynamics in Patients With Atherosclerotic Intracranial Arterial Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10688
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2019-06

CONDITIONS: Atherosclerosis
Keywords: Atherosclerotic Intracranial Arterial Stenosis; Intensive Rosuvastatin Therapy; Computed Tomography Perfusion (CTP)
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard dose (Active Comparator): Drug: Rosuvastatin rosuvastatin 10 mg daily for 52 weeks.
  Interventions: Drug: Rosuvastatin
- intensive dose (Experimental): Drug: Rosuvastatin rosuvastatin 20 mg daily for 52 weeks.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — standard or intensive dose rosuvastatin therapy based on other routine medication for stroke for 52 weeks.
  Other Names: Crestor

SUMMARY:
Atherosclerotic intracranial arterial stenosis (AICAS) corresponds to luminal narrowing of the major intracranial arteries. The prevalence of intracranial atherosclerotic stenosis accounts for 33% to 67% of stroke or transient ischemic attack (TIA) cases in China and other countries in Asia. AICAS is also highly associated with the risk of stroke recurrence. Possible mechanisms of cerebral infarction secondary to AICAS are likely linked with hemodynamic compromise distal to site of stenosis.

Computed tomography perfusion (CTP) can be used to evaluate vasoreactivity and cerebrovascular reserve in patients with AICAS and predict future stroke. The parameters of CTP include ①cerebral blood flow(CBF),② cerebral blood volume(CBV) and ③mean transit time(MTT). Relative regional cerebral blood flow (rCBF) was evaluated as the percentage radioisotope counts in the region of interest (ROI) of the affected side against the corresponding ROI in the unaffected contralateral side.

Statins can decrease the incidence of transient ischemic attack or ischemic stroke and improve stroke outcome. Few studies focus on the relationship between statins therapy and cerebral perfusion.

Whether intensive rosuvastatin therapy compared with standard rosuvastatin therapy can improve hemodynamic situation and cerebral perfusion status in AICAS has not been illustrated.

Based on those studies, the investigators hypothesized that intensive rosuvastatin may also improve the symptoms of AICAS not only through enhancing the stability of atherosclerotic plaques, but also its pleiotropic effects. So it can change the hemodynamic status around the plaque and increase cerebral flow in the downstream territory. So in this study the investigators try to analysis statin's impact on the hemodynamic changes as well as the downstream perfusion which is determined by CTP.

DETAILED DESCRIPTION:
This is an prospective, randomized, single-blind, single center clinical trial to evaluate the effect of intensive rosuvastatin therapy compared with standard rosuvastatin therapy on improve the cerebral perfusion in Chinese patients with atherosclerotic intracranial arterial stenosis between 50-99%.

The study will enroll 44 patients and randomly divided into 2 groups: standard dose rosuvastatin therapy (SRT 10mg/day)and intensive dose rosuvastatin therapy (IRT 20mg/day)in a 1:1 ratio. Both groups will be prescribed with statin based on other routine medication for stroke for 52 weeks. CTP will be performed at baseline and 52 weeks after treatment. Lipid levels and biochemical examinations will be obtained at baseline and 13, 26, 39, 52 week. AEs(Adverse Events)/SAEs(Serious Adverse Events) will be collected and recorded in CRF(Case Report Form) from the signing of informed consent throughout the study until and including the last visit.

Study Endpoints: Primary endpoint: Compared with standard dose rosuvastatin therapy 10mg/day, the change of relative cerebral blood flow (CBF) by CTP after intensive dose rosuvastatin therapy 20mg/day treatment for 52 weeks.Secondary endpoints: (1) Compared with standard dose rosuvastatin therapy 10mg/day, the changes of relative cerebral blood volume (CBV) by CTP after rosuvastatin 20mg/d treatment for 52 weeks (2) Compared with standard dose rosuvastatin therapy 10mg/day, the changes of relative mean transit time (MTT) by CTP after rosuvastatin 20mg/d treatment for 52 weeks (3) Compared with standard dose rosuvastatin therapy 10mg/day, the changes of lipid parameters (LDL-C, HDL-C, TG(Triglyceride), TC(Total Cholesterol), Apo A and Apo B ) after rosuvastatin 20mg/d for 52 weeks (4) Safety.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Male and female adults aged 18-80years old
3. Recent (within 3 months) ischemic stroke or TIA;
4. Intracranial large artery (intracranial internal artery, middle cerebral artery M1, vertebral artery and basilar artery) stenosis between 50-99%.
5. Statin naïve:defined as receiving no statin therapy within 3 months

Exclusion Criteria:

1. Cardioembolic stroke;
2. Rosuvastatin use is contraindicated;
3. Allergic to contrast agents;
4. Chronic devastating illness, multiple organ failure;
5. Dementia or mental disorder unable to return for repeat brain CTP.
6. Administration of lipid-lowering drugs (statin, clofibrate, probucol or analog, nicotinic acid, or other prohibited drug) before enrollment.
7. Active liver disease or aminopherase ≧3 ULN(Upper Limit of Normal)
8. Renal function damage. GFR（Glomerular Filtration Rate） ﹤30ml/min

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
the change of relative cerebral blood flow (CBF) （ml/100g/min）by CTP | 52 weeks

SECONDARY OUTCOMES:
the changes of relative cerebral blood volume (CBV)（ml/100g） by CTP | 52 weeks
the changes of relative mean transit time (MTT)（min） by CTP | 52 weeks
the changes of lipid parameters (LDL-C,mmol/L；HDL-C,mmol/L；TG,mmol/L；TC,mmol/L；Apo A，mmol/L；Apo B，mmol/L ) | 13, 26, 39, 52 week
myopathic events, hepatic function, renal function and other adverse events. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, Ph.D, Principal Investigator — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China